CLINICAL TRIAL: NCT00697918
Title: An Extension Study to Evaluate the Safety and Effectiveness of RWJ-333369 as Adjunctive Therapy in Korean and Japanese Patients With Partial Onset Seizures
Brief Title: Long Term Effectiveness and Safety Study for RWJ-333369 as Adjunctive Therapy in Korean and Japanese Patients With Partial Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014287; 333369-KJ-03
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Seizures
Keywords: Partial onset seizure; Adjunctive therapy
MeSH Terms: conditions — Seizures | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

ARMS (1):
- 001 (Experimental): RWJ-333369100 mg to 400 mg twice daily
  Interventions: Drug: RWJ-333369

INTERVENTIONS:
Drug: RWJ-333369 — 100 mg to 400 mg twice daily

SUMMARY:
The purpose of this study is to evaluate the long-term safety of RWJ-333369 at doses between 200-800 mg/day in Korean and Japanese patients who have completed the preceding study (333369-KJ-02).

DETAILED DESCRIPTION:
Despite the introduction of new antiepileptic drugs into overseas clinical settings after 1990's, there still exist those patients who cannot control seizures, and thus the advent of newer antiepileptic drugs is being desired. This is a multicenter, open-label, extension study in patients who have completed the preceding study (333369-KJ-02) and scheduled to continue until the study drug is approved. This study consists of Period 1 (1 year) and Period 2 (only in Japan; planned to continue until the drug is approved Primary objective of this study is to evaluate the long-term safety (Adverse event, Lab test, Electrocardiogram, Vital signs, Pregnancy test, Physician Withdrawal Checklist) of RWJ-333369 at doses between 200-800 mg/day in patients who have completed the preceding study. Secondary objective of this study is to evaluate the long-term effectiveness of RWJ-333369 at doses between 200-800 mg/day in patients who have completed the preceding study. Period 1:RWJ-333369 will be started at 400 mg/day. RWJ-333369 100 mg tablets or 200 mg tablets will be orally administered with noncarbonated water twice daily. The dose will be adjusted between 200 mg/day and 800 mg/day based on effectiveness and tolerance. Period 2: The dose will be adjusted between 200 mg/day and 800 mg/day based on effectiveness and tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the preceding study (333369-KJ-02) who have completed Double-Blind Treatment Phase of preceding study

Exclusion Criteria:

* Considered ineligible as study patients by the investigator

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Adverse events (subjective/objective findings), blood pressure, pulse rate, body temperature, weight, 12-lead ECG, laboratory tests, pregnancy test. Time measure is 1 year. | For 1 year.

SECONDARY OUTCOMES:
Percent reduction in partial seizure frequency | For 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.